CLINICAL TRIAL: NCT05412563
Title: Exploring The Role Of Palliative Care In Phase 1 Enrolled Pediatric Oncology Patients
Status: Terminated | Type: Observational
Why Stopped: IRB approval to Close to accrual on 2-18-2025: Thematic saturation reached and enrolling further participants was deemed not necessary.
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EPCP1; NCI-2022-04886 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Quality of Life
Keywords: Palliative Care; Pediatric Oncology Patients; Caregiver; Phase I studies; Associated Distress; Hopes; Worries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is being conducted to learn more about the patient/family experience when opting to enroll in Phase I clinical trials and their quality of life (QOL) while receiving experimental therapy. Palliative care (PC) has the potential to be beneficial for these families and further studies are needed to determine the most effective way for integration of PC into the care of patients enrolled on experimental clinical trials.

Primary Objective

* To qualitatively assess the patient and family experience, their hopes and worries and associated distress while deciding to enroll on a Phase I clinical trial.

DETAILED DESCRIPTION:
Eligible Parent Research Participants (PRPs) who consent will participate in one audio recorded interview in which they are asked about 8-10 questions. The interview can be conducted in person, over the phone, or WebEx/Zoom (audio only). The interview will last about 30 to 60 minutes. PRPs can opt to complete interviews immediately or at a scheduled date that is convenient to the PRP.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver is 18 years of age or older
* Caregiver is related to the patient in one of the following ways: biological parent, stepparent, or primary legal guardian
* If more than 1 set of parents are involved in the patient's care (e.g., 2 biologic and 2 stepparents or partners) involved, the caregiver with legal decision- making responsibilities will be eligible for participation
* Caregiver is comfortable speaking and reading English

Exclusion Criteria:

* Those who do not meet inclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Those who meet the Inclusion criteria and consent to participate
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Qualitative assessment of patient and family experience | Up to approximately 8 months after enrollment
  Qualitative analysis of interviews done with parents of children with cancer who are enrolling in phase 1 studies will be performed. Broad thematic domains will be identified through a rigorous review of transcript data, with the development of codes to delineate conceptual categories. Domains will be further sub-stratified as text analysis progresses in order to identify new themes and formulate new concepts and theories. To enhance construct validity and reliability of identified domains, data will be audited by an expert panel of PPC investigators with proficiency in communication-based research, including both clinicians and researchers. Coding schemata will remain flexible to accommodate expansion of the list as the PI and expert panel agree on new code additions. Following the well-described processes of disassembling and reassembling coding categories, emerging themes will be categorized and refined, with the ultimate goal of theory-building.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Kaye, MD, MPH, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - National Cancer Institute/National Institutes of Health, Bethesda, Maryland
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols